CLINICAL TRIAL: NCT00552344
Title: A Phase IIIb, Multinational, Open-label, follow-on Trial to C87085 Designed to Assess the Long-term Safety of Certolizumab Pegol, a Pegylated Fab' Fragment of a Humanized Anti-TNF-alpha Monoclonal Antibody, Administered at Weeks 0, 2 and 4, and Then Every 4 Weeks Thereafter, in Subjects With Moderately to Severely Active Crohn's Disease Who Have Participated in Study C87085
Brief Title: A Study to Evaluate Safety of Long Term Therapy of Certolizumab Pegol Patients With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87088; 2007-002716-26 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2016-01

CONDITIONS: Crohn Disease
Keywords: CDP 870; Certolizumab Pegol; CIMZIA; Crohn's Disease; Crohn Disease; CD Induction; Induction; Clinical response; Clinical remission
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): Certolizumab Pegol 200 mg/vial; 400 mg subcutaneously at Week 0, 2 and 4, thereafter 400 mg subcutaneously at every 4 weeks.
  Interventions: Biological: Cimzia

INTERVENTIONS:
Biological: Cimzia — * Active substance: Certolizumab Pegol
  * Pharmaceutical form:first reconstituted, lyophilized powder formulation of CZP and after implementation of Amendment 2 (after 401 subjects were enrolled) prefilled syringe
  * Concentration: 200 mg/ml
  * Route of Administration: Subcutaneous use
  Other Names: Certolizumab Pegol; CDP870; CZP

SUMMARY:
The primary objective of the study is to assess the safety of long term therapy with Certolizumab Pegol in those subjects participating in study C87085 [NCT00552058].

DETAILED DESCRIPTION:
This study consisted of:

* Induction Period (dosing at Weeks 0, 2, and 4)
* Maintenance Dosing (dosing every 4 weeks up to Week 260)
* End of Treatment Visit that occurred at Week 262/Withdrawal Visit and a Safety Follow-up Visit (SFU; 12 weeks after final dose)

ELIGIBILITY:
Inclusion Criteria:

* Subject participated in study C87085 [NCT00552058] in which the subject completed the study at Week 6
* Subject is capable of providing informed consent, which must be obtained prior to any study related procedures
* Have a chest X-ray taken at Visit 1 that is read by a qualified radiologist or pulmonary physician, with no evidence of current active Tuberculosis (TB) or old inactive TB
* Subject has taken a TB survey and is committed to comply with TB prophylaxis if applicable

Exclusion Criteria:

* Subject is experiencing an ongoing serious adverse event assessed as being related to study medication or is experiencing a serious adverse event that is still not assessable
* Subject has an intercurrent illness that requires termination of treatment, such as a serious infection (e.g. TB, pneumonia, sepsis, pyelonephritis, fistula abscess)
* Subject is non-compliant with TB prophylactic treatment (if applicable)
* Subject has had a chest X-ray at Visit 1 that shows an abnormality suggestive of a malignancy or active infection, including TB
* Female who is pregnant or breast feeding
* Female of child bearing age or post puberty males not practicing effective birth control
* Subject is expecting to receive any live virus or bacterial vaccination within 3 months of first Study Medication administration, during the trial or 3 months after last dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2008-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (100):
- United States (20):
  - 284, Lakewood, Colorado
  - 285, Littleton, Colorado
  - 278, New Port Richey, Florida
  - 300, Winter Park, Florida
  - 276, Chicago, Illinois
  - 279, Louisville, Kentucky
  - 275, Metairie, Louisiana
  - 307, Monroe, Louisiana
  - 281, Annapolis, Maryland
  - 295, Towson, Maryland
  - 310, Chesterfield, Michigan
  - 298, Rochester, Minnesota
  - 272, Raleigh, North Carolina
  - 296, Cincinnati, Ohio
  - 289, Cleveland, Ohio
  - 280, Lancaster, Pennsylvania
  - 305, Germantown, Tennessee
  - 306, Germantown, Tennessee
  - 308, Norfolk, Virginia
  - 290, Seattle, Washington
- Australia (8):
  - 15, Concord, New South Wales
  - 20, Box Hill, Victoria
  - 12, Footscray, Victoria
  - 16, Parkville, Victoria
  - 14, Bankstown
  - 11, Fitzroy
  - 13, Fremantle
  - 18, Garran
- 270, Vienna, Austria
- Belgium (5):
  - 32, Bonheiden
  - 31, Ghent
  - 35, Leuven
  - 34, Liège
  - 30, Roeselare
- Brazil (6):
  - 52, Porto Alegre, Rio Grande do Sul
  - 45, Belo Horizonte
  - 41, Curitiba
  - 51, Rio de Janeiro
  - 53, Santos
  - 55, São Paulo
- Canada (8):
  - 64, Edmonton, Alberta
  - 60, Winnepeg, Manitoba
  - 67, Hamilton, Ontario
  - 62, Kingston, Ontario
  - 63, London, Ontario
  - 70, London, Ontario
  - 66, Toronto, Ontario
  - 68, Toronto, Ontario
- Czechia (3):
  - 95, Hradec Králové
  - 97, Hradek Kralove
  - 98, Prague
- Estonia (2):
  - 100, Tallinn
  - 101, Tartu
- Germany (4):
  - 140, Homburg
  - 137, Kiel
  - 144, Ulm
  - 130, Wilhelmshaven
- Hungary (7):
  - 151, Budapest
  - 155, Budapest
  - 156, Budapest
  - 154, Győr
  - 150, Nagykanizsa
  - 153, Szeged
  - 152, Szombathely
- Israel (7):
  - 161, Beersheba
  - 164, Haifa
  - 167, Holon
  - 163, Kfar Saba
  - 166, Petha Tikva
  - 160, Tel Aviv
  - 169, Ẕerifin
- Italy (3):
  - 176, Padua
  - 171, Roma
  - 174, Roma
- Latvia (3):
  - 191, Riga
  - 192, Riga
  - 193, Riga
- New Zealand (5):
  - 202, Milford, Auckland
  - 204, Newton, Wellington Region
  - 201, Auckland
  - 200, Christchurch
  - 203, Hamilton
- Poland (6):
  - 217, Częstochowa
  - 218, Częstochowa
  - 210, Lodz
  - 211, Warsaw
  - 212, Warsaw
  - 213, Wroclaw
- Romania (2):
  - 221, Cluj-Napoca
  - 225, Constanța
- Russia (4):
  - 232, Kazan'
  - 230, Moscow
  - 234, Moscow
  - 233, Saint Petersburg
- Ukraine (6):
  - 258, Dniepropetrovsk
  - 251, Donetsk
  - 256, Kiev
  - 259, Kiev
  - 257, Lviv
  - 254, Simferopol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in May 2008 and concluded in Dec 2014. Participant Flow refers to the Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Pre-assignment Details: 406 subjects were screened: 3 subjects were considered as screen failures and were not enrolled. 403 subjects entered the study from C87085. 1 subject was enrolled in this study, but did not receive any open-label study medication and was withdrawn from the study; this subject was, therefore, not included in any of the analyses.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 402
Completed | 87
Not Completed | 315
Not completed — Lack of Efficacy | 55
Not completed — Loss of efficacy | 75
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 48
Not completed — SAE, non-fatal | 6
Not completed — AE, non-serious non-fatal | 38
Not completed — SAE,non-fatal+AE,non-serious non-fatal | 62
Not completed — SAE, fatal + AE, non-serious non-fatal | 1
Not completed — Other Reason | 22

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication. Demographics presented below were collected at Screening of the feeder study C87085.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
Age, Customized [Number; unit: Participants]
  18 - < 65 years | 393
  65 - < 85 years | 9
  >= 85 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221
  Male | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) During the Duration of the Study C87088 (up to 272 Weeks)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From study start to the end of the Safety Follow-up Period (up to 272 weeks)
Population: Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 89.6

2. Primary Outcome: Percentage of Subjects With at Least One Serious Adverse Event (SAE) During the Duration of the Study C87088 (up to 272 Weeks)
Description: An SAE is defined as any untoward medical occurrence that occurs at any dose which results in death, is life threatening, requires hospitalization, results in persistent/significant disability/incapacity, is an infection that requires parenteral antibiotics, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From study start to the end of the Safety Follow-up Period (up to 272 weeks)
Population: Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 37.1

3. Secondary Outcome: Percentage of Subjects Achieving Harvey Bradshaw Index (HBI) Remission (HBI ≤ 4) at Study Completion Visit (Week 262)
Description: HBI remission is defined as total HBI score of 4 points or less. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well being. The first three parameters are scored for the previous day.
Time Frame: Week 262
Population: Intention-to-Treat (ITT) population including all enrolled subjects irrespective of any protocol deviations who received at least 1 open-label injection of study treatment and who had at least 1 efficacy measurement after the first open-label injection.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Certolizumab Pegol (Intention-to-Treat): Certolizumab Pegol 200 mg/vial; 400 mg subcutaneously at Week 0, 2 and 4, thereafter 400 mg subcutaneously at every 4 weeks.
  The ITT Population includes all enrolled subjects irrespective of any protocol deviations who received at least 1 open-label injection of study treatment and who had at least 1 efficacy measurement after the first open-label injection.
Arm/Group | Certolizumab Pegol (Intention-to-Treat)
Number analyzed (Participants) | 397
percentage of subjects | 11.6 [8.4 to 14.7]

4. Secondary Outcome: Percentage of Subjects Achieving Inflamatory Bowel Disease Questionnaire (IBDQ) Remission (IBDQ ≥ 170) at Study Completion Visit (Week 262)
Description: IBDQ remission is defined as having a total IBDQ score of 170 points or greater. IBDQ score consists of 32 questions eaching having a score of 1 to 7. Overall scores range from 32 to 224.
Time Frame: Week 262
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol (Intention-to-Treat)
Number analyzed (Participants) | 397
percentage of subjects | 7.8 [5.2 to 10.4]

5. Secondary Outcome: Plasma Concentration of Certolizumab Pegol After 1 Year (Week 52)
Description: Plasma samples for determination of Certolizumab Pegol were taken prior to Certolizumab Pegol administration.
Time Frame: Week 52
Population: Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
μg/mL | 6.317 [5.407 to 7.381]

6. Secondary Outcome: Percentage of Subjects With Positive Anti-CZP Anti-body Status at Any Time From Week 0 of the Feeder Study C87085 to the Study Completion Visit in C87088
Description: Subjects are counted as antibody positive to Certolizumab Pegol if they have at least one positive result from Week 0 in the previous study C87085 [NCT00552058] to the Last Visit in this study. A positive result is defined as Anti-CZP antibody levels > 2.4 units/mL.
Time Frame: From Week 0 of study C87085 [NCT00552058] to Study Completion Visit (Week 262) of C87088 (up to 268 weeks)
Population: Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 402
percentage of subjects | 10.2

ADVERSE EVENTS:
Time Frame: Adverse Events presented below where collected from the Final Visit in Feeder study C87085 (Week 0) over the whole study period until the Safety-Follow-Up Visit (up to 274 weeks).
Description: Adverse Events refer to the Safety Population including all enrolled subjects who received at least 1 open-label injection of study medication.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 149/402
Other Adverse Events (participants affected / at risk) | 351/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=402)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Anal fistula (Gastrointestinal disorders) | 2 (3)
Anorectal disorder (Gastrointestinal disorders) | 1 (1)
Colon dysplasia (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 51 (59)
Enteritis (Gastrointestinal disorders) | 1 (1)
Enterocolonic fistula (Gastrointestinal disorders) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (2)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileal fistula (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 11 (11)
Intestinal perforation (Gastrointestinal disorders) | 2 (2)
Intestinal stenosis (Gastrointestinal disorders) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (6)
Subileus (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1)
Mass (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Unevaluable event (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 4 (4)
Abdominal sepsis (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 2 (2)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Psoas abscess (Infections and infestations) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Vulval abscess (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
Investigation (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (5)
Syncope (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Acute psychosis (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Depression suicidal (Psychiatric disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 5 (5)
Renal colic (Renal and urinary disorders) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Physical assault (Social circumstances) | 1 (1)
Social stay hospitalisation (Social circumstances) | 1 (1)
Victim of abuse (Social circumstances) | 1 (1)
Arteritis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=402)
Anaemia (Blood and lymphatic system disorders) | 34 (45)
Crohn's disease (Gastrointestinal disorders) | 127 (191)
Abdominal pain (Gastrointestinal disorders) | 75 (122)
Diarrhoea (Gastrointestinal disorders) | 61 (93)
Nausea (Gastrointestinal disorders) | 46 (63)
Vomiting (Gastrointestinal disorders) | 43 (60)
Dyspepsia (Gastrointestinal disorders) | 32 (37)
Abdominal pain upper (Gastrointestinal disorders) | 24 (28)
Pyrexia (General disorders) | 54 (106)
Influenza like illness (General disorders) | 23 (40)
Upper respiratory tract infection (Infections and infestations) | 63 (99)
Nasopharyngitis (Infections and infestations) | 46 (88)
Influenza (Infections and infestations) | 30 (35)
Sinusitis (Infections and infestations) | 29 (48)
Urinary tract infection (Infections and infestations) | 25 (31)
Bronchitis (Infections and infestations) | 21 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 (79)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (40)
Headache (Nervous system disorders) | 45 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (49)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (27)
Rash (Skin and subcutaneous tissue disorders) | 27 (39)
Hypertension (Vascular disorders) | 28 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days